CLINICAL TRIAL: NCT01223612
Title: Diabetic Macula Oedema. A Prospective Randomised Study Comparing the Detailed Functional and Anatomical Changes of Repeated Pan Anti-VEGF Therapy With Ranibizumab Versus Conventional Macular Laser Therapy.
Brief Title: Lucentis (Ranibizumab) in Diabetic Macular Oedema: a Treatment Evaluation
Acronym: LUCIDATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYKP1015
Record Dates: First submitted 2010-10-18; First posted 2010-10-19 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes Mellitus; Diabetes Complications; Retinal Diseases; Edema; Endothelial Growth Factors; Monoclonal Antibodies; Ranibizumab; Laser therapy
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Diabetes Complications; Retinal Diseases; Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranibizumab (Experimental): Intravitreal injection of ranibizumab
  Interventions: Drug: Ranibizumab
- Laser (Active Comparator): Modified ETDRS laser
  Interventions: Procedure: Modified ETDRS laser

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injection of 0.5mg in 0.05ml. One injection at baseline, 4 and 8 weeks then four-weekly as required to 44 weeks.
  Other Names: Lucentis
  Arms: Ranibizumab
Procedure: Modified ETDRS laser — Argon laser therapy to the macula in accordance with the modified ETDRS protocol at baseline, 12, 24 and 36 weeks.
  Other Names: Argon laser photocoagulation
  Arms: Laser

SUMMARY:
This exploratory study will compare the effects of ranibizumab treatment with conventional macular laser therapy for patients with diabetic macular oedema.

The study hypothesises that treatment with ranibizumab may be superior to laser treatment in terms of improving vision and decreasing retinal thickness.

Patients will be randomised to receive either repeated injections of ranibizumab every 4 weeks for 48 weeks or macular laser therapy every 12 weeks for 48 weeks.

At baseline, and then at 12, 24 and 48 weeks, patients will undergo detailed testing to provide information on the structure and function of the retina with both of these treatments.

DETAILED DESCRIPTION:
Adult patients with centre-involving diabetic macular oedema will be recruited to this single-centre study. Patients will undergo detailed baseline evaluation which will include:

* vision testing
* optical coherence tomography scanning
* fundus fluorescein angiography
* microperimetry
* colour contrast sensitivity testing
* electrophysiological testing

Patients will be randomised 2:1 to receive either ranibizumab intravitreal injection 4-weekly for 48 weeks or modified ETDRS macular laser therapy 12-weekly for 48 weeks.

Both groups of patients will return at 12, 24 and 48 weeks for repeat testing of the parameters evaluated at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2)
* Retinal thickening due to diabetic macular oedema involving the centre of the macula and OCT central subfield ≥ 300 microns
* Best corrected visual acuity in the study eye between 55 and 79 ETDRS letters at 1 metre (Snellen equivalent ≥ 6/24 and ≤ 6/9)
* Media clarity, pupillary dilation, and subject cooperation sufficient for adequate fundus photographs
* Intraocular pressure less than 30 mmHg
* Ability to return for study visits
* Visual acuity in fellow eye ≥ 2/60
* Fellow eye has received no anti-VEGF treatment within the past 3 months and no expectation of such treatment in next 12 months
* No previous laser within 3 months of randomisation
* Ability to give informed consent throughout the duration of the study

Exclusion Criteria:

* Macular ischaemia
* Macular oedema from a cause other than diabetic macular oedema
* Co-existent ocular disease
* Presence of an ocular condition such that visual acuity would not improve from resolution of macular oedema
* Presence of an ocular condition that might affect macular oedema or alter visual acuity during the course of the study
* A substantial cataract that is likely to be decreasing visual acuity by 3 lines or more
* History of treatment for diabetic macular oedema at any time in the past 3 months
* History of panretinal scatter photocoagulation (PRP) within 3 months prior to randomisation
* Anticipated need for PRP in the 6 months following randomisation.
* Proliferative diabetic retinopathy in the study eye.
* A condition that, in the opinion of the investigator, would preclude participation in the study.
* Haemoglobin A1c > 11.0 %
* A past medical history of significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant
* Blood pressure >170/100 mmHg
* Myocardial infarction, other cardiac event requiring hospitalisation, stroke, transient ischaemic attack, or treatment for acute congestive heart failure within 6 months prior to randomisation
* Major surgery within 28 days prior to randomisation or major surgery planned during the next 12 months at baseline
* Participation in an investigational trial within 30 days of randomisation that involved treatment with any drug that has not received regulatory approval at the time of study entry. Note: subjects cannot receive another investigational drug while participating in the study
* Systemic anti-VEGF or pro-VEGF treatment within 3 months prior to randomisation
* Pregnant or lactating women or women intending to become pregnant within the study period including 3 months after study cessation
* History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery) within prior 3 months or anticipated within the next 6 months following randomisation.
* Aphakia
* Uncontrolled glaucoma
* External ocular infection, including conjunctivitis, chalazion, or severe blepharitis
* Known allergy to fluorescein dye or to any component of the study drug
* Fertile male unwilling to use contraception for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Functional and anatomical change in the retina | 48 weeks
  This is an exploratory study. The primary outcome measure is the change in retinal function and anatomy at 48 weeks compared to baseline, as assessed by fluorescein angiography, microperimetry and electrophysiological testing.

SECONDARY OUTCOMES:
Mean ETDRS acuity | 48 weeks
  Difference in mean ETDRS visual acuity between the two study arms.
OCT macular thickness | 48 weeks
  Difference in mean OCT central retinal thickness between the two study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Philip G Hykin, FRCS FRCOphth, Principal Investigator — Moorfields Eye Hospital NHS Trust
Locations (1):
- Moorfields Eye Hospital, London, United Kingdom